CLINICAL TRIAL: NCT03750526
Title: Investigate the Effectiveness of Augmented Reality and Repetitive Transcranial Magnetic Stimulation Technology in Persons With Stroke
Brief Title: Effectiveness of Augmented Reality and Repetitive Transcranial Magnetic Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Lai chien hung, Professor, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201703084
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Stroke
Keywords: Repetitive transcranial magnetic stimulation (rTMS); Augmented reality (AR); stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- rTMS and AR group (Experimental): Ten participants in group A will undergo repetitive transcranial magnetic stimulation (real, 1 Hz, 15 minutes), follow by a session of augmented reality exercise (45 minutes), 3 days per week for 4 weeks.
  Interventions: Behavioral: rTMS and AR
- Sham rTMS and AR group (Active Comparator): Ten participants in group B will receive repetitive transcranial magnetic stimulation (sham,1 Hz, 15 minutes), follow by a session of augmented reality exercise (45 minutes), 3 days per week for 4 weeks.
  Interventions: Behavioral: Sham rTMS and AR
- AR group (Active Comparator): Ten participants in group C will undergo augmented reality exercise 60 minutes a day and 3 days per week for four weeks.
  Interventions: Behavioral: AR
- Conventional physiotherapy group (Active Comparator): Ten participants allocated to the group D will receive conventional physiotherapy 60 minutes a day and 3 days per week for four weeks.
  Interventions: Behavioral: Conventional physiotherapy

INTERVENTIONS:
Behavioral: rTMS and AR — rTMS performs 1Hz,15 minutes real rTMS. AR intervention contains weight-shift exercise, strengthening of lower limb and balance training for 45 minutes.
  Arms: rTMS and AR group
Behavioral: Sham rTMS and AR — Sham rTMS applies 1Hz, 15 minutes sham rTMS. AR intervention includes weight-shift exercise, strengthening of lower limb and balance training for 45 minutes.
  Arms: Sham rTMS and AR group
Behavioral: AR — AR intervention contains weight-shift exercise, strengthening of lower limb and balance training for 60 minutes.
  Arms: AR group
Behavioral: Conventional physiotherapy — Conventional physiotherapy includes rolling, sitting, balance exercise, standing, overground walking, facilitation of the paretic limbs, and so on for 60 minutes.
  Arms: Conventional physiotherapy group

SUMMARY:
This study is to investigate the combined effects of repetitive Transcranial Magnetic Stimulation (rTMS) and Augmented Reality (AR) intervention on cortical excitability, balance, gait, activity in individuals with stroke. Forty participants will be recruited in this study. They will be allocated to four group: rTMS and AR group (10), sham rTMS and AR group (10), AR group (10), and conventional physiotherapy group (10).

DETAILED DESCRIPTION:
Participants will be randomized allocated to four groups: rTMS and AR group, sham rTMS and AR group, AR group ,and conventional physiotherapy group in current study. All participants underwent four weeks, 3 sessions per week, and 60 minutes per session training program. Motor evoked potential (MEP), Time up go test (TUG), Berg Balance Scale (BBS), Fugl-Meyer Assessment (FMA), Multi-directional Reach Test (MDRT),The Postural Assessment Scale for Stroke Patients (PASS), and Taiwanese Depression Questionnaires (TDQ) will be assessed before and after intervention in all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Cognitive ability is sufficient to understand the nature of study (Mini-Mental State Examination score was above 23).
2. Participants suffer from unilateral hemiplegia caused by a first-ever stroke.
3. Participants are stable in medical and psychological condition.

Exclusion Criteria:

1. Participants have other neurologic problems that can affect balance and walking ability.
2. Participants take of drugs or have other medical condition that can affect balance and function.
3. Participants have contraindications for rTMS intervention such as pacemaker, cochlear implants, metal in the brain or skull, open wound of brain, or history of epilepsy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of Time Up Go test (TUG) | Measurement before and after intervention ( week 0 and at the end of week 4) in four groups
  The TUG test will ask participants to stand up, walk for 3 m, turn, walk back and sit down as fast as they can during the test, and the time requires for each patient to complete the test is recorded.

SECONDARY OUTCOMES:
Change of Berg Balance Scale (BBS) | Measurement before and after intervention ( week 0 and at the end of week 4) in four groups
  Participants performed a series of 14 functional balance tasks, including maintaining a quiet stance, sitting-to-standing, shifting weight and reaching, turning in place, standing on one leg, and maintaining a tandem stance. Each task was scored on a 5-point ordinal scale (from 0 to 4). A score of 0 denotes the inability of the participant to perform the task, and a score of 4 denotes that the participant can complete the task based on a preset criterion. The highest possible score is 56.
Change of Motor evoked potential (MEP) | Measurement before and after intervention ( week 0 and at the end of week 4) in four groups
  Motor evoked potential (MEP) is recorded from tibialis anterior muscles following direct transcranial magnetic stimulation (TMS) of motor cortex. All TMS is delivered with the participant seated upright on the chair. Both passive and active conditions, participants are instructed to relax their right leg in the seated position. TMS is delivered over the motor cortex (M1) using a concave double cone coil (Magstim Co., United Kingdom) attached to a BiStim magnetic stimulator (Magstim Co., United Kingdom). To locate the optimal site, stimuli are delivered over various points along the M1. The optimal site is the location on the M1 that evoked the greatest MEP amplitude in the bilateral tibialis anterior muscles. The onset latency and onset to peak amplitude will be assessed.
Change of Fugl-Meyer Assessment (FMA)-Lower extremity | Measurement before and after intervention ( week 0 and at the end of week 4) in four groups
  Fugl-Meyer Assessment-Lower extremity is used to measure lower-limb recovery in stroke rehabilitation studies.The scale has 6 items ranging from reflex activity to voluntary motor control. Each item further comprises components, with a total of 17. Scoring is done on a 3-point ordinal scale ranges from 0 (no performance) to 2 (faultless performance). The total score range from 0 (no motor function) to 34 (good motor recovery).
Change of Multi-directional Reach Test (MDRT) | Measurement before and after intervention ( week 0 and at the end of week 4) in four groups
  Participants will be required to reach in the forward, left and right directions. The test is performed with the participant in standing. It is the measure of the difference, in centimeters, between arm's length with arms at 90° flexion/ abduction and maximal forward, left and right directions reaching respectively, using a fixed base of support. The test uses a centimeters measuring device against a wall at shoulder height.
Change of The Postural Assessment Scale for Stroke Patients (PASS) | Measurement before and after intervention ( week 0 and at the end of week 4) in four groups
  The Postural Assessment Scale for Stroke Patients (PASS) is a postural assessment scale specifically designed to assess and monitor postural control after stroke. It contains 12 four-level items of varying difficulty for assessing ability to maintain or change a given lying, sitting, or standing posture. The PASS consists of 2 sections with a 4-point scale to describe each task. The total score ranges from 0 - 36. A score of 0 denotes the inability of the participant to perform the task, and a score of 3 denotes that the participant can complete the task based on a preset criterion. The highest possible score is 36.
Change of Taiwanese Depression Questionnaires (TDQ) | Measurement before and after intervention ( week 0 and at the end of week 4) in four groups
  Taiwanese Depression Questionnaires (TDQ) contains 18 items to screen the situation of depression within a week. The TDQ, which is a 4-point scale with 18 items, is a culturally specific depression self-rating instrument for effective screening of depression in Taiwan and has satisfactory reliability and validity. Subjects are guided to rate each item on a scale from 0 to 3 on the basis of "how often you felt the physical and emotional aspects during the past week". Zero denotes never, three means always. TDQ scores range from 0 to 54.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hung Lai, MD PhD, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical university Hospital, Taipei, Taiwan